CLINICAL TRIAL: NCT07201220
Title: The Effect of Relaxation Meditation During the First Stage of Labor on Childbirth Self-Efficacy and Fear in Primiparous Women: A Randomized Controlled Trial
Brief Title: Meditation in Early Labor: Impact on Self-Efficacy and Childbirth Fear in First-Time Mothers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seyhan District Health Directorate, Adana (Other)
Responsible Party: Principal Investigator, EMEL SALCAN, PHD Midwife, Seyhan District Health Directorate, Adana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022.03.06/123
Record Dates: First submitted 2025-09-09; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Meditation
MeSH Terms: interventions — Meditation

STUDY DESIGN:
Intervention Model Description: After informing the pregnant women about the study and the procedures to be implemented, informed consent will be obtained from those who agree to participate. Following this, participants will complete the data collection form, and pre-test questionnaires will be administered. Subsequently, relaxation meditation will be played via headphones during labor, and the questionnaires will be applied again as post-tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A Randomized Controlled Experimental Study (Experimental): Experimental Group:
  30 primiparous women in the first stage of labor receive relaxation meditation during labor. Pre- and post-tests using the Childbirth Self-Efficacy Inventory Short Form and W-DEQ Version A are applied. Data collected between 01.04.2025 and 01.08.2025 at a tertiary hospital in Turkey.
  Control Group:
  30 primiparous women in the first stage of labor receive standard care without intervention. The same pre- and post-tests are applied. Data collected in the same period and setting.
  Interventions: Behavioral: meditation

INTERVENTIONS:
Behavioral: meditation — The study is planned to include 60 pregnant women (30 in the experimental group and 30 in the control group) in the first stage of labor. After informing the participants about the study and obtaining informed consent, pre-test scales will be administered. Relaxation meditation will be applied during labor for the experimental group, followed by post-test scales.

SUMMARY:
Aim-Introduction:

The feeling of uncertainty about what will happen during labor, and the mother's perception of inadequacy regarding childbirth, can lead to anxiety and stress in some pregnant women, resulting in fear of childbirth and avoidance behaviors. This study was conducted to examine whether there are significant differences in childbirth self-efficacy and fear of childbirth between primiparous pregnant women who practiced meditation and those who did not during the first stage of labor.

Materials and Methods:

This experimental study is planned to be conducted between 01.04.2025 and 01.08.2025 with a total of 60 pregnant women (30 in the experimental group and 30 in the control group) who applied to the delivery unit of a tertiary hospital in Turkey and were in the first stage of labor. After informing the pregnant women about the study and the procedures to be implemented, written informed consent was obtained from those who agreed to participate. Subsequently, the pre-tests of the relevant scales and the data collection form were administered. The relaxation meditation during childbirth was applied to the experimental group, followed by the post-tests of the same scales.

Data were collected using the "Childbirth Self-Efficacy Inventory Short Form" and the "Wijma Delivery Expectancy/Experience Questionnaire (W-DEQ) Version A." Descriptive statistics and hypothesis tests will be used for data analysis.

DETAILED DESCRIPTION:
Introduction:

This study aims to examine whether there are significant differences in childbirth self-efficacy and fear of childbirth between primiparous pregnant women who practice meditation (experimental group) and those who do not (control group) during the first stage of labor. Childbirth is a physiological process for every woman, but feelings of uncertainty, perceived inadequacy, anxiety, and stress can lead to fear of childbirth and avoidance behavior. Studies show that 6.3-75% of pregnant women experience fear of childbirth, with 6-10% affected severely. This fear can be influenced by biological, psychological, social, and secondary factors such as previous traumatic experiences or negative birth stories. Furthermore, gestational age and parity also play important roles in the emergence of birth fear.

Fear of childbirth can result in complications such as prolonged labor, emergency or elective cesarean delivery, postpartum depression, post-traumatic stress disorder, and disruption in mother-infant bonding. Various methods, including cognitive-behavioral techniques, psychoeducation, and relaxation therapies like hypnobirthing, are used to manage this fear. Research suggests that birth fear is not solely linked to pain or information deficits but to many other factors, including a woman's sense of self-efficacy.

Self-efficacy refers to a person's belief in their ability to complete tasks or overcome challenges. A woman with high self-efficacy is more likely to manage stress-inducing situations, such as labor, by trusting her own capabilities. Increasing self-efficacy and reducing fear of childbirth can be achieved through relaxation techniques, one of which is meditation. Meditation involves mental training that helps individuals find strength and solutions to problems, promoting relaxation that may alleviate both mental and physical tension. During pregnancy and labor, meditation can assist in reducing anxiety and enhancing positive birth experiences.

Aim:

The study aims to investigate whether relaxation through meditation in the first stage of labor can enhance self-efficacy and reduce fear of childbirth in primiparous women, contributing to a less stressful and anxious labor process. Gestational age and parity are known to influence childbirth fear. The research will evaluate whether meditation can help reduce anxiety and foster self-efficacy, aiding in a more manageable birth experience.

Research Problem:

Does a significant difference exist between the self-efficacy and fear of childbirth of primiparous women who receive meditation during the first stage of labor and those who do not?

Keywords: Primiparous pregnancy, Meditation, Childbirth Self-Efficacy, Fear of Childbirth.

ELIGIBILITY:
Inclusion Criteria:

Primiparous pregnant women

In the first stage of labor

Singleton pregnancy

Aged 18 and above

Able to provide informed consent

No high-risk pregnancy or psychiatric diagnosis

Exclusion Criteria:

Multiparous women

High-risk pregnancy

Previous experience with meditation during labor

Communication difficulties

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in perceived childbirth self-efficacy measured by the Childbirth Self-Efficacy Inventory Short Form (CBSEI-SF) | From the beginning of the active phase of the first stage of labor to 1 hour after the intervention
  Perceived childbirth self-efficacy is assessed using the Childbirth Self-Efficacy Inventory Short Form (CBSEI-SF). The scale is administered during the active phase of the first stage of labor (before the intervention), and re-administered 1 hour after relaxation meditation. Change in scores indicates the effect of the intervention on participants' self-efficacy levels.

SECONDARY OUTCOMES:
Change in fear of childbirth measured by the Wijma Delivery Expectancy/Experience Questionnaire Version A (W-DEQ Version A) | From the beginning of the active phase of the first stage of labor to 1 hour after the intervention
  Fear of childbirth is assessed using the Wijma Delivery Expectancy/Experience Questionnaire Version A (W-DEQ Version A). The scale is applied before the relaxation meditation during the active phase of the first stage of labor and re-applied 1 hour after the intervention. The change in scores reflects the effect of the intervention on fear of childbirth.intervention and re-administered within 24 hours after delivery to evaluate changes in fear levels among participants.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Seyhan İlçe Sağlık Müdürlüğü, Adana, Adana
  - Seyhan İlçe Sağlık Müdürlüğü, Seyhan, Adana